CLINICAL TRIAL: NCT03921996
Title: Extended Pelvic Lymph Node Dissection vs. no Pelvic Lymph Node Dissection at Radical Prostatectomy for intermediate-and High-risk Prostate Cancer: An International, Multicenter, Randomized Phase III Trial
Brief Title: Extended Pelvic Lymph Node Dissection vs. no Pelvic Lymph Node Dissection at Radical Prostatectomy for intermediate-and High-risk Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to lack of funding.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 09/18
Record Dates: First submitted 2019-04-18; First posted 2019-04-19 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Extended pelvic lymph node dissection; Pelvic lymph node dissection; ePLND; Prostate Cancer; intermediate prostate cancer; High-risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: SAKK 09/18 is an international, multicenter, randomized, phase III surgical intervention trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A: ePLND (Experimental): Radical prostatectomy with extended pelvic lymph node dissection
  Interventions: Procedure: Radical prostatectomy (RP) followed by ePLND
- arm B: no PLND (Active Comparator): Radical prostatectomy only
  Interventions: Procedure: Radical prostatectomy (RP) only

INTERVENTIONS:
Procedure: Radical prostatectomy (RP) followed by ePLND — ePLND is performed either before or after radical prostatectomy and includes the removal of all nodal and fibro-fatty tissue
  Arms: arm A: ePLND
Procedure: Radical prostatectomy (RP) only — Radical prostatectomy
  Arms: arm B: no PLND

SUMMARY:
For patients with intermediate-risk prostate cancer plus a predicted risk of >5% for positive lymph nodes and with high-risk prostate cancer, international guidelines recommend ePLND along with the RP. Besides an improved accuracy in staging, the therapeutic role of ePLND remains controversial. We hypothesize that ePLND prolongs time to biochemical recurrence (BCR) and prostate cancer-specific survival (PCSS) in intermediate- and high-risk PCa patients.

DETAILED DESCRIPTION:
Radical prostatectomy (RP) is the surgical standard treatment for men with localized prostate cancer (PCa) and a life expectancy of > 10 years. RP is a treatment option for localized PCa that shows benefit in prostate cancer-specific survival (PCSS) and overall survival compared to conservative management. According to the guideline recommendations of the European Association of Urology (EAU), RP should be accompanied by extended pelvic lymph node dissection (ePLND) in patients with intermediate-risk PCa (D'Amico classification) and > 5% nomogram (Briganti) predicted risk of positive lymph nodes and in all high-risk PCa cases.

Besides an improved accuracy in staging, the therapeutic role of ePLND remains controversial. The primary goal of this trial is to provide high-level evidence regarding the therapeutic benefit of ePLND in intermediate- and high-risk PCa patients without clinical evidence of nodal involvement. It is hypothesized that ePLND prolongs time to biochemical recurrence (BCR) and prostate cancer-specific survival (PCSS) in intermediate- and high-risk PCa patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures.
* Histologically proven localized adenocarcinoma of the prostate.
* High-risk prostate cancer or intermediate-risk prostate cancer defined by D'Amico classification system, with an estimated risk of >5% of lymph node metastasis.
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence.
* Age ≥ 18 years and ≤ 80 years.
* WHO performance status 0-1.
* Adequate condition (ASA ≤ III) for general anesthesia and radical prostatectomy surgery.
* Baseline Quality of Life (QoL) questionnaires have been completed.

Exclusion criteria

* Any pre-operative evidence for T4 disease.
* Metastatic prostate cancer according to staging or evidence of lymph node metastasis by imaging, defined as any pelvic lymph node >9 mm in the short axis or positive lymph nodes detected by imaging techniques with sensitivities similar or better than PSMA-PET or Choline-PET prior to surgery.
* PSA ≥ 50 ng/ml.
* Any prior neo-adjuvant, local or systemic treatment for prostate cancer (alpha reductase inhibitors for treatment of benign hyperplasia are allowed)
* Previous pelvic lymph node dissection.
* Any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Time to biochemical recurrence (BCR) | From the date of randomization until the date of biochemical recurrence, assessed up to 15 years after surgery
  The primary endpoint of this trial is time to BCR, defined as time from randomization to biochemical recurrence, defined as serum PSA level ≥ 0.2 ng/ml, with a second confirmatory serum PSA level ≥ 0.2 ng/ml. Patients not experiencing an event will be censored at the date of the last available assessment or at the start of adjuvant or salvage treatment, if any.

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) persistence | From the date of surgery to 14 weeks after surgery
  PSA persistence is defined as failure to reach a PSA value of <0.1 ng/ml within 12 weeks (+ 2 weeks) postoperatively.
  Patients with no assessments within the first 12 weeks (+ 2 weeks) after surgery will be counted as failures for this endpoint
Time to initiation of adjuvant or salvage therapies | From the date of randomization until the date of start of any type of adjuvant or salvage therapy, assessed up to 15 years after surgery
  Time to initiation of adjuvant or salvage therapies will be calculated as the time from randomization to the start of any type of adjuvant or salvage therapy. Patients not starting adjuvant or salvage therapies are censored at the last date they were known to be alive.
Time to loco-regional recurrence | From the date of randomization until the date of local or regional recurrence, assessed up to 15 years after surgery
  Time to loco-regional recurrence will be calculated from randomization until local (prostate bed) or regional (extent of ePLND template) recurrence, whichever occurs first. Patients not experiencing an event will be censored at the date of the last available assessment or at the start of adjuvant or salvage therapy, if any.
Time to distant metastasis | From the date of randomization until the date of first occurrence of distant metastasis, assessed up to 15 years after surgery
  Time to distant metastasis will be calculated from randomization until first occurrence of distant metastasis. Patients not experiencing an event will be censored at the date of the last available assessment.
Prostate cancer-specific survival (PCSS) | From the date of randomization until the date of death due to prostate cancer, assessed up to 15 years after surgery
  PCSS will be calculated as the time from randomization to the date of death due to prostate cancer. Patients who died due to other reasons will be censored at the time of death. All other patients will be censored at the last date they were known to be alive.
  Causes of death may require critical review by the coordinating investigator and the medical advisor. Particular attention will be paid to men who have been reported as having died from prostate cancer without previously reported progression or recurrence and men who were reported as having died from non-prostate cancer causes after developing biochemical or clinical progression.
Overall survival (OS) | From the date of randomization until the date of death, assessed up to 15 years after surgery
  OS will be calculated from randomization until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
Intraoperative complications | During surgery
  Intraoperative complications will be assessed using the CLASSIC system.
Postoperative complications | From the date of surgery to 14 weeks after surgery
  Postoperative complications will be assessed using the Clavien-Dindo classification.
Adverse events (AE) | From the date of registration to 15 years after surgery
  AEs will be assessed according to NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrill A. Rentsch, MD-PhD, Study Chair — University Hospital Basel, Department of Urology
Locations (11):
- Switzerland (11):
  - Kantonsspital Aarau AG, Aarau
  - Universitätsspital Basel, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux Universitaires Genève, Geneva
  - Kantonsspital Baselland, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Spital Thurgau AG (Frauenfeld and Münsterlingen), Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich
  - Universitätsspital Zürich, Zurich